CLINICAL TRIAL: NCT06585774
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Axatilimab and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease (AXemplify-357)
Brief Title: A Study to Evaluate Axatilimab and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease
Acronym: AXemplify-357
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCA34176-357; 2023-510292-65-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05544032 (Available)
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; Adrenal Cortex Hormones; Prednisone; Methylprednisolone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axatilimab + Corticosteroids (Experimental): Axatilimab and Corticosteroids at the protocol-defined dose.
  Interventions: Drug: INCA034176; Drug: Corticosteroids
- Placebo + Corticosteroids (Experimental): Matching placebo and Corticosteroids at the protocol-defined dose.
  Interventions: Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Drug: INCA034176 — IV infusion
  Other Names: Axatilimab
  Arms: Axatilimab + Corticosteroids
Drug: Placebo — IV infusion
  Arms: Placebo + Corticosteroids
Drug: Corticosteroids — Oral/IV Infusion
  Other Names: prednisone, methylprednisolone, prednisolone

SUMMARY:
This study will be conducted to compare the efficacy of axatilimab versus placebo in combination with corticosteroids as initial treatment for moderate or severe chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years of age at the time of informed consent.
* New-onset moderate or severe cGVHD, as defined by the 2014 NIH Consensus Development Project Criteria for Clinical Trials in cGVHD, requiring systemic therapy.
* History of allo-HCT from any donor HLA type (related or unrelated donor with any degree of HLA matching) using any graft source (bone marrow, peripheral blood stem cells, or cord blood). Recipients of myeloablative, nonmyeloablative, or reduced-intensity conditioning are eligible.
* Adequate hematologic function with ANC ≥ 0.5 × 109/L independent of growth factors for at least 7 days prior to study entry.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Received more than 1 prior allo-HCT. Prior autologous HCT is allowed.
* Has overlap cGVHD, defined as simultaneous presence of features or characteristics of aGVHD in a patient with cGVHD.
* Received more than 7 days of systemic corticosteroid treatment for cGVHD or unable to begin a prednisone dose ≥ 1.0 mg/kg per day (or methylprednisolone equivalent) for cGVHD.
* Received previous systemic treatment for cGVHD, including extracorporeal photopheresis.
* Systemic treatment with CNIs or mTOR inhibitors started within 2 weeks prior to C1D1.
* Prior treatment with CSF-1R targeted therapies.
* Active, uncontrolled bacterial, fungal, parasitic, or viral infection.
* Evidence of relapse of the primary hematologic disease or treatment for relapse after the allo-HCT was performed, including DLIs for the treatment of molecular relapse.
* History of acute or chronic pancreatitis.
* Active symptomatic myositis.
* History or current diagnosis of cardiac disease indicating significant risk of safety for participation in the study, such as uncontrolled or significant cardiac disease.
* Severe renal impairment, that is, estimated CrCl < 30 mL/min measured or calculated by Cockcroft-Gault equation in adults and Schwartz formula in pediatric participants, or endstage renal disease on dialysis.
* Impaired liver function, defined as total bilirubin > 1.5 × ULN and/or ALT and AST > 3 × ULN in participants with no evidence of liver cGVHD.
* Pregnant or breastfeeding.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | Up to 3 years
  Defined from the date of randomization to the date of any predefined event, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response (OR) | 6 months
  Defined for each treatment group as CR or PR at 6 months Cycle 7 (28-day cycles), Day 1, in the absence of new systemic therapy for cGVHD. Responses defined by the 2014 NIH consensus criteria.
Event Free Survival 2 | Up to 3 years
  Defined from the date of randomization to the date of any predefined event, whichever occurs first.
Proportion of participants with a ≥ 7-point improvement in mLSS total score | Up to 3 years
Overall Response | 12 Months
  Defined as CR or PR at 12 months in the absence of new systemic therapy for cGVHD.
DOR (in responders only) | Up to 3 years
  Defined as the time from the date of first response (PR or CR) to the date of progression of cGVHD from nadir in any organ, start of new systemic treatment for cGVHD, or death from any cause, whichever comes first.
Best Overall Response (BOR) | Up to 3 years
  Defined as the best response of CR or PR at any timepoint up to the initiation of new therapy for cGVHD.
Overall Survival (OS) | Up to 3 years
  Defined as the time from the date of randomization to the date of death due to any cause.
Nonrelapse mortality (NRM) | Up to 3 years
  Defined as the time from the date of randomization to the date of death in the absence of primary hematologic disease relapse.
Failure-free survival (FFS) | Up to 3 years
  Defined as the time from the date of randomization to the date of addition or initiation of another systemic therapy for cGVHD, relapse of underlying disease, or death due to any cause.
Relapse of hematologic diseases | Up to 3 years
  Defined as the reappearance of symptoms of underlying disease.
Time to primary hematologic disease relapse | Up to 3 years
  Defined as the time from the date of randomization to the date of relapse.
Percent reduction in daily corticosteroid dose | 6 months
Proportion of participants who tapered off all corticosteroids | 6 months
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 3 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Change from baseline in circulating monocyte number and phenotype (CD14/16) | Up to 3 years and 30 days
Change from baseline in soluble markers for bone resorption and formation, including bone-specific alkaline phosphatase (BAP) and C-terminal telopeptide (CTX) | Up to 3 years and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation
Locations (113):
- United States (29):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute Downtown Orlando, Orlando, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Hematology Oncology, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Transplant Institute, San Antonio, Texas
  - Intermountain Blood and Marrow Transplant, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - West Virginia University Cancer Institute, Morgantown, West Virginia
- Australia (3):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health Medical Oncology and Clinical Haematology, Heidelberg, Victoria
- Austria (5):
  - Landeskrankenhaus Universitatsklinikum Graz, Graz
  - Innsbruck University Hospital, Innsbruck
  - Ordensklinikum Linz Gmbh Elisabethinen, LINZ CET
  - Akh Und Medizinische Universitat Wien Universitatsklinik Fur Innere Medizin I, Vienna
  - St. Anna Childrens Hospital, Vienna
- Canada (7):
  - Alberta'S Children Hospital, Calgary, Alberta
  - Bc Children'S Hospital, Vancouver, British Columbia
  - Queen Elizabeth Ii Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hospital Maisonneuve Rosemont, Montreal, Quebec
  - Vancouver General Hospital, Vancouver
- Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Chu Amiens Picardie - Hopital Sud, Amiens
  - Hopitaux de Brabois, Nancy
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Chu de Nice - Hospital L Archet, Nice
  - Hospital Saint Louis, Paris
  - Hospital Saint Antoine, Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
- Germany (13):
  - University Medical Center Rwth Aachen, Aachen
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Bonn, University Hospital Bonn, Bonn
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - University Hospital Duesseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Halle (Saale), Halle
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Klinikum Der Philipps-Universitaet Marburg, Marburg
  - Universitatsklinikum Munster, Münster
- St. James Hospital, Dublin, Ireland
- Italy (15):
  - Azienda Ospedaliero-Universitaria Di Alessandria Ss.Antonio E Biagio E Cesare Arrigo, Alessandria
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Asst Degli Spedali Civili Di Brescia, Brescia
  - Irccs Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Raffaele - Milano, Milan
  - Azienda Ospedaliera Di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Irccs Fondazione Policlinico San Matteo, Pavia
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - Azienda Policlinico Umberto 1 Universita Sapienza Di Roma, Rome
  - Ospedale Pediatrico Bambino Gesu Irccs, Rome
  - I.R.C.C.S. Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Card. G. Panico, Tricase
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (13):
  - Anjo Kosei Hospital, Aichi
  - Fujita Health University Hospital, Aichi
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Kobe City Medical Center General Hospital, Hyōgo
  - Tokai University Hospital, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Gunma Saiseikai Maebashi Hospital, Maebashi
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo Hokkaido
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
- Amsterdam University Medical Centre, Amsterdam, Netherlands
- Spain (10):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Institut Catala Doncologia Ico - Hospital Duran I Reynals Location, L'Hospitalet de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - Bristol Haematology and Oncology Centre, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Marsden Hospital, London
  - University College London Hospitals (Uclh), London
  - Manchester University Nhs Foundation Trust, Manchester
  - Nottingham University Hospitals, Nottingham
  - Plymouth Hospitals Nhs Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to evaluate Axatilimab and Corticosteroids as Initial Treatment for Chronic Graft-Versus-Host Disease — https://incyteclinicaltrials.com/studies/inca34176-357